CLINICAL TRIAL: NCT02561689
Title: SEALANT-DK: Longevity and Efficacy of 6 Resin Sealants Used for Sealing Permanent Teeth in Children and Adolescents
Acronym: SEALANT-DK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Azam Bakhshandeh, Associate professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCopenhagen
Record Dates: First submitted 2014-12-02; First posted 2015-09-28 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Dental Caries
Keywords: Occlusal caries; Resin fissure sealant; Longevity; Effectiveness
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fissure sealant material 1 (Experimental): Fissure sealing with Delton FS+ Fissure sealing withClinpro Sealant Fissure sealing withGrandio Seal Fissure sealing withControl Seal Fissure sealing withUltraSeal XT+ UltraSeal XT hydro
  Interventions: Other: Fissure sealing
- Fissure sealant material 2 (Experimental): Fissure sealing with Delton FS+ Fissure sealing withClinpro Sealant Fissure sealing withGrandio Seal Fissure sealing withControl Seal Fissure sealing withUltraSeal XT+ UltraSeal XT hydro
  Interventions: Other: Fissure sealing

INTERVENTIONS:
Other: Fissure sealing — Procedure:
  * The included teeth of the participating patients will in any case be sealed, but in this study, the operator is not free to choose the material, the material choice is determined by randomisation
  * Standardized radiographs (bitewings) will be taken before treatment and after 1, 2, 3 years and possibly after 5 years. Baseline radiograph can be taken up to six months before treatment. If using conventional radiography, double-film packs will be used. A maximum of 8/10 bitewings will be taken during the study period of 3/5 years
  * The occlusal surface is sealed by the dentist or dental hygienist.
  * Clinical evaluation of the quality of sealants and the need for re-treatments during the follow-up will be performed after 1, 2 and 3 years and possibly after 5 years

SUMMARY:
Background: Occlusal caries is the main reason for restorative therapy in the young permanent dentition, but restorations have limited survival time and may also weaken the tooth. An intact fissure sealing is an effective preventive treatment of occlusal caries lesions and may be used therapeutically to arrest the caries progression. However, the major challenge with fissure sealants is the frequent need for re-treatments, mostly due to inadequate retention.

Purpose: To quantify the longevity and effectiveness of the 6 resin sealants used prophylactically and therapeutically in permanent molar teeth.

Study design: The study is carried out as a prospective, clinically controlled study with split-mouth design, where each of the 60 dentists/dental hygienists from 13 municipalities in Denmark uses 2 of the 6 sealants. The treatments are examined clinically and radiologically after 1, 2, 3, and 5 years.

DETAILED DESCRIPTION:
The choice of the two materials is randomized and carried out so that all materials are used equally frequent and with an even distribution between dentists and dental hygienists.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents 5-14 years of age
* Children with 2, 4, 6 or 8 molars assessed to be in need of prophylactic or therapeutic sealing
* The radiographic penetration of the occlusal caries lesion must be limited halfway through the dentin

Exclusion Criteria:

* In case the occlusal surface is restored with communication between the restoration and the included lesion
* Subjects with chronic diseases that could affect their caries pattern
* Pain in teeth

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 248 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Longevity of 6 resin fissure sealants assessed by defined scoring system | 5 years
  Clinical scoring system: 1: Intact sealing (success), 2: Partly loss of sealant (failure); 3: Total loss of sealant (failure)
Efficacy of 6 resin fissure sealants assessed by defined radiological scoring system | 5 years
  Radiographic scoring system: 1:Regression in depth of lesion (success), 2: Unchanged depth of lesion (success); 3: Progression in depth of lesion (failure)

CONTACTS AND LOCATIONS:
Overall Officials: Azam AB Bakhshandeh, PhD, Study Chair — University of Copenhagen; Vibeke VQ Qvist, Dr Odont, Study Chair — University of Copenhagen
Locations (1):
- Dental Health Care in Denmark, Copenhagen, Denmark